CLINICAL TRIAL: NCT01688596
Title: Infiltration of Bupivacaine Local Anesthetic to Trocar Insertion Sites After Laparoscopic Hysterectomy: A Randomized, Double-Blind, Placebo-Controlled Trial
Brief Title: Injection of Local Anesthetic to Trocar Insertion Sites After Laparoscopy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Matthew Davies, Professor, Division of Urogynecology and Minimally Invasive GYN Surgery, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 40708
Record Dates: First submitted 2012-09-07; First posted 2012-09-20 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2018-03

CONDITIONS: Pain, Postoperative
Keywords: Local; Anesthesia; Pain; Laparoscopic hysterectomy; Trocar site; Port site
MeSH Terms: conditions — Pain, Postoperative; Pain | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Treatment (No Intervention): The "No Treatment" group includes patients undergoing laparoscopic hysterectomy without local infiltration of bupivacaine.
- Bupivacaine (Active Comparator): The "Bupivacaine Arm" includes all patients who will receive bupivacaine injection on their trocar sites after the laparoscopic hysterectomy is completed. Bupivacaine (0.25%) will be injected through the closed incisions ensuring subcutaneous tissue, fascia, muscle and pre-peritoneal space of the trocar incision sites are infiltrated. All incisions 8 mm and greater are injected with 10 cc while all incisions 5 mm or less are infiltrated with 5 cc.
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine (0.25%) will be injected through the closed trocar incisions after completion of the laparoscopic hysterectomy case.
  Other Names: Marcaine
  Arms: Bupivacaine

SUMMARY:
The primary objective of this study is to assess if injection of local anesthetic to the laparoscopic trocar sites after a hysterectomy will make a difference in a patient's pain after surgery.

DETAILED DESCRIPTION:
The growing interest in minimally invasive gynecologic surgeries have increased the number of patients undergoing laparoscopic hysterectomies. Although many patients are being discharged home the same day of surgery, majority of patients complain of immediate postoperative pain after a laparoscopic hysterectomy. Since postoperative pain is usually transient and improves over a short period of time, infiltration of local anesthetic to trocar insertion sites might alleviate the patient's discomfort during the recovery period. Immediate post-operative pain relief further facilitates early discharge and faster patient recovery.

Published data regarding the effects of preemptive port site local anesthesia in gynecologic operative laparoscopy have been limited and controversial. Visceral pain control through afferent nerve block could minimize pain perception especially during the first postoperative hours. This study aims to assess the influence of infiltration of local anesthetic to trocar insertion sites after laparoscopic hysterectomy on postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled for a laparoscopic hysterectomy for benign indications at the Department of Obstetrics & Gynecology's Division of Minimally Invasive Surgery at Milton S. Hershey Medical Center will be included.

Exclusion Criteria:

* Patients who are scheduled for a hysterectomy through the vaginal or abdominal approach will be excluded. Patients with preoperative indications of endometriosis or chronic pelvic pain will also be excluded since these patients could potentially have higher thresholds of pain.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Harkins, MD, Study Director — Milton S. Hershey Medical Center; Maria Teresa Tam, MD, Principal Investigator — Milton S. Hershey Medical Center; Matthew Davies, MD, Study Chair — Milton S. Hershey Medical Center
Locations (1):
- Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Einarsson JI, Sun J, Orav J, Young AE. Local analgesia in laparoscopy: a randomized trial. Obstet Gynecol. 2004 Dec;104(6):1335-9. doi: 10.1097/01.AOG.0000146283.90934.fd. PMID 15572499
- [Background] Kim JH, Lee YS, Shin HW, Chang MS, Park YC, Kim WY. Effect of administration of ketorolac and local anaesthetic infiltration for pain relief after laparoscopic-assisted vaginal hysterectomy. J Int Med Res. 2005 Jul-Aug;33(4):372-8. doi: 10.1177/147323000503300402. PMID 16104440
- [Background] Saleh A, Fox G, Felemban A, Guerra C, Tulandi T. Effects of local bupivacaine instillation on pain after laparoscopy. J Am Assoc Gynecol Laparosc. 2001 May;8(2):203-6. doi: 10.1016/s1074-3804(05)60578-6. PMID 11342725
- [Background] Ghezzi F, Cromi A, Bergamini V, Raffaelli R, Crotti S, Segredini R, Bolis P. Preemptive port site local anesthesia in gynecologic laparoscopy: a randomized, controlled trial. J Minim Invasive Gynecol. 2005 May-Jun;12(3):210-5. doi: 10.1016/j.jmig.2005.03.007. PMID 15922977
- [Background] Marks JL, Ata B, Tulandi T. Systematic review and metaanalysis of intraperitoneal instillation of local anesthetics for reduction of pain after gynecologic laparoscopy. J Minim Invasive Gynecol. 2012 Sep-Oct;19(5):545-53. doi: 10.1016/j.jmig.2012.04.002. Epub 2012 Jul 3. PMID 22763313
- [Background] Chou YJ, Ou YC, Lan KC, Jawan B, Chang SY, Kung FT. Preemptive analgesia installation during gynecologic laparoscopy: a randomized trial. J Minim Invasive Gynecol. 2005 Jul-Aug;12(4):330-5. doi: 10.1016/j.jmig.2005.05.005. PMID 16036193
- [Background] Fong SY, Pavy TJ, Yeo ST, Paech MJ, Gurrin LC. Assessment of wound infiltration with bupivacaine in women undergoing day-case gynecological laparoscopy. Reg Anesth Pain Med. 2001 Mar-Apr;26(2):131-6. doi: 10.1053/rapm.2001.21836. PMID 11251136
- [Background] Ke RW, Portera SG, Bagous W, Lincoln SR. A randomized, double-blinded trial of preemptive analgesia in laparoscopy. Obstet Gynecol. 1998 Dec;92(6):972-5. doi: 10.1016/s0029-7844(98)00303-2. PMID 9840560
- [Background] Salman MA, Yucebas ME, Coskun F, Aypar U. Day-case laparoscopy: a comparison of prophylactic opioid, NSAID or local anesthesia for postoperative analgesia. Acta Anaesthesiol Scand. 2000 May;44(5):536-42. doi: 10.1034/j.1399-6576.2000.00508.x. PMID 10786738
- [Background] Goldstein A, Grimault P, Henique A, Keller M, Fortin A, Darai E. Preventing postoperative pain by local anesthetic instillation after laparoscopic gynecologic surgery: a placebo-controlled comparison of bupivacaine and ropivacaine. Anesth Analg. 2000 Aug;91(2):403-7. doi: 10.1097/00000539-200008000-00032. PMID 10910857

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing laparoscopic surgery at Penn State Milton S. Hershey Medical Center were recruited between 3/13 and 6/13. Allocated to CPP or no CPP based on usual clinical definitions.
Pre-assignment Details: Patients in each group (Chronic Pelvic Pain and No Chronic Pelvic Pain) were randomized to receive either a bupivacaine block at each trocar site or no block. Standardization of amount of local block received was based on trocar size of 5mm or less vs. 8mm and or greater.
Period: Overall Study
Arm/Group | No Treatment | Bupivacaine
Started | 67 | 68
Completed | 59 | 59
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Treatment | Bupivacaine | Total
Number analyzed (Participants) | 67 | 68 | 135
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 67 | 68 | 135
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.3 (8.4) | 38.6 (10.5) | 38.5 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 68 | 135
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 67 | 68 | 135
Parity [Count of Participants; unit: Participants] | 67 | 68 | 135
Chronic Pelvic Pain [Number; unit: participants] | 36 | 35 | 71

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Pain Score Evaluated by Numerical Rating Scale (NRS)
Description: Postoperative pain is measured on day of surgery after trocar incisions are closed and injected with local anesthetic. Postoperative pain is evaluated with the Numerical Rating Scale (NRS) at 4 hrs after the surgery. The Numerical Rating Scale is a scale from 0 to 10 that measures pain severity, where 0 equates to "no pain" and 10 equates to "unable to move".
Time Frame: 4 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Treatment | Bupivacaine
Number analyzed (Participants) | 65 | 59
units on a scale | 4.1 (2.4) | 3.4 (2.6)

2. Primary Outcome: Postoperative Pain Score
Description: Postoperative pain is measured on day of surgery after trocar incisions are closed and injected with local anesthetic. Postoperative pain is evaluated with the Numerical Rating Scale (NRS) at 6 hrs after the surgery. The Numerical Rating Scale is a scale from 0 to 10 that measures pain severity, where 0 equates to "no pain" and 10 equates to "unable to move".
Time Frame: 6 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Treatment | Bupivacaine
Number analyzed (Participants) | 43 | 40
units on a scale | 4.7 (2.3) | 4.3 (2.1)

3. Primary Outcome: Postoperative Pain Score
Description: Postoperative pain is measured on day of surgery after trocar incisions are closed and injected with local anesthetic. Postoperative pain is evaluated with the Numerical Rating Scale (NRS) at 24 hrs after the surgery. The Numerical Rating Scale is a scale from 0 to 10 that measures pain severity, where 0 equates to "no pain" and 10 equates to "unable to move".
Time Frame: 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | No Treatment | Bupivacaine
Number analyzed (Participants) | 29 | 28
units on a scale | 3.5 (2.4) | 4.0 (1.8)

4. Secondary Outcome: Estimated Blood Loss > 200 mL
Description: Estimated blood loss will be measured in (mL) on the day of surgery after completing the procedure. Blood loss will be categorized as >200 mL vs. <= 200 mL.
Time Frame: day of surgery after procedure completion
Measure: Count of Participants; unit: Participants
Arm/Group | No Treatment | Bupivacaine
Number analyzed (Participants) | 67 | 67
Participants | 2 | 2

5. Secondary Outcome: Surgical Complications
Description: Intraoperative complications include injury to bowel, bladder, blood vessels, nerves and hemorrhage. Perioperative complications include urinary tract infections, urinary retention, ileus, myocardial infarction, atrial fibrillation, pulmonary edema, atelectasis, pneumonia, renal and cerebrovascular morbidity, thromboembolic complications (DVT and PE). Postoperative complications include pulmonary, renal, and cerebrovascular morbidity, wound and vaginal vault complications (infection, separation, and dehiscence), septicemia, thromboembolic events, and re-operation.
Time Frame: From date of randomization up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | No Treatment | Bupivacaine
Number analyzed (Participants) | 67 | 68
Participants | 0 | 0

6. Secondary Outcome: Operating Time
Description: Operating time measured in minutes
Time Frame: start to end of patient's surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | No Treatment | Bupivacaine
Number analyzed (Participants) | 67 | 67
minutes | 73.3 (33.9) | 63.8 (24.5)

7. Secondary Outcome: Length of Hospital Stay >= 24 Hours
Description: Length of hospital stay will be measured on the day of surgery after completing the procedure to when the patient is discharged from the hospital. Length of stay will be categorized as less than 24 hours vs. greater than or equal to 24 hours.
Time Frame: from time surgery completed to time patient discharged
Measure: Count of Participants; unit: Participants
Arm/Group | No Treatment | Bupivacaine
Number analyzed (Participants) | 67 | 67
Participants | 36 | 30

8. Secondary Outcome: Histopathologic Diagnosis
Description: Histopathologic diagnosis describes the findings seen on tissue pathology and microscopy and is defined as one of the following: endometriosis, leiomyoma, adenomyosis, or other.
Time Frame: Histopathologic diagnosis will be measured on the day of surgery after completing the procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | No Treatment | Bupivacaine
Number analyzed (Participants) | 67 | 67
Participants
  Endometriosis | 26 | 21
  Leiomyoma | 10 | 12
  Adenomyosis | 5 | 3
  Other | 26 | 31

9. Other Pre Specified Outcome: Primary Surgical Finding
Description: The primary intra-operative finding found during surgery, defined as one of the following: endometriosis, pelvic adhesive disease, leiomyoma, or other.
Time Frame: Surgical findings will be measured on the day of surgery after completing the procedure.
Measure: Count of Participants; unit: Participants
Arm/Group | No Treatment | Bupivacaine
Number analyzed (Participants) | 67 | 67
Participants
  Endometriosis | 37 | 41
  Pelvic adhesive disease | 12 | 5
  Leiomyoma | 6 | 9
  Other | 12 | 12

ADVERSE EVENTS:
Arm/Group | No Treatment | Bupivacaine
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/68
Other Adverse Events (participants affected / at risk) | 0/67 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No